CLINICAL TRIAL: NCT03395184
Title: A PHASE 2A, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, PARALLEL GROUP STUDY TO EVALUATE THE EFFICACY AND SAFETY OF ORAL PF-06651600 AND PF-06700841 AS INDUCTION AND OPEN LABEL EXTENSION TREATMENT IN SUBJECTS WITH MODERATE TO SEVERE CROHN'S DISEASE
Brief Title: Study To Evaluate The Efficacy And Safety Of Oral PF-06651600 And PF-06700841 In Subjects With Moderate To Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7981007; 2017-003359-43 (EudraCT Number); PIZZICATO (Other: Alias Study Number)
Record Dates: First submitted 2017-12-05; First posted 2018-01-10 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — PF-06651600; PF-06700841

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06700841 or placebo (Experimental)
  Interventions: Drug: Placebo PF-06700841; Drug: PF-06700841
- PF-06651600 or placebo (Experimental)
  Interventions: Drug: PF-06651600 Placebo; Drug: PF-06651600

INTERVENTIONS:
Drug: PF-06651600 Placebo — 12 weeks, followed by PF-06651600, 50 mg once daily (QD) for 52 weeks
  Arms: PF-06651600 or placebo
Drug: PF-06651600 — 200 mg QD for 8 weeks, followed by 50 mg QD up to 56 weeks
  Arms: PF-06651600 or placebo
Drug: Placebo PF-06700841 — 12 weeks, followed by PF-06700841, 30 mg QD for 52 weeks
  Arms: PF-06700841 or placebo
Drug: PF-06700841 — 60 mg QD for 12 weeks followed by 30 mg QD for up to 52 weeks
  Arms: PF-06700841 or placebo

SUMMARY:
The objectives of this study are to evaluate the efficacy, safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-06651600 (200 mg for 8 weeks followed by 50 mg for 4 weeks) dosed once daily and PF-06700841 (60 mg for 12 weeks) dosed once daily during an induction period of 12 weeks, followed by an open label extension period at doses of 50 mg and 30 mg of PF 06651600 and PF 06700841, respectively, for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and/or female subjects 18 years to 75 years of age
2. Documented diagnosis of ileal, ileocolonic, or colonic CD with a minimum disease duration of 3 months, as determined by endoscopic and histopathology assessment.
3. Endoscopic confirmation of active disease with total SES CD total score of at least 7. For isolated ileal disease, SES CD total score should be at least 4.
4. An average daily liquid/soft stool frequency (SF) greater than or equal to 2.5 or daily abdominal pain (AP) greater than or equal to 2.0.
5. Must have inadequate response to, loss of response to, or intolerance to at least one conventional therapy for CD:

   •Steroids; Immunosuppressants (azathioprine [AZA], 6 MP, or methotrexate [MTX]); Anti TNF inhibitors (infliximab, adalimumab,certolizumab); Anti integrin inhibitors (eg, vedolizumab); Anti IL 12/23 inhibitor (ustekinumab).
6. Subjects currently receiving the following treatment for CD are eligible providing they have been on stable doses as described below:

   * Oral corticosteroids (prednisone or equivalent up to 25 mg/day; budesonide up to 9 mg/day). Stable dose for at least 2 weeks prior to baseline. If oral corticosteroids have been recently discontinued, they must have been stopped at least 2 weeks prior to baseline. Decreases in steroid use due to AEs are allowed.
   * Oral 5 ASA or sulfasalazine are allowed providing that the dose is stable for at least 4 weeks prior to baseline.
   * Crohn's disease related antibiotics are allowed providing that the dose is stable for at least 4 weeks prior to baseline. If antibiotics are stopped prior to baseline, they must be discontinued at least 4 days prior to baseline.

Exclusion Criteria:

1. Diagnosis of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, radiation colitis, diverticular disease, ulcerative colitis (UC), or clinical findings suggestive of UC.
2. Presence of active (draining) fistulae or intra abdominal or perineal abscesses.
3. Strictures with obstructive symptoms.
4. Short bowel syndrome.
5. History of bowel perforation requiring surgical intervention within the past 12 months.
6. Previous bowel surgery resulting in an existing stoma. Subjects who have a j pouch are excluded, as a j pouch can result in a stoma.
7. History of bowel surgery within 6 months prior to baseline.
8. Subjects displaying clinical signs of fulminant colitis or toxic megacolon.
9. Subjects with primary sclerosing cholangitis.
10. Subjects with evidence of colonic adenomas, dysplasia or neoplasia.
11. Abnormal findings on the chest x ray film such as presence of tuberculosis (TB), general infections, heart failure, or malignancy.
12. Any history of either untreated or inadequately treated latent or active TB infection, current treatment for active or latent TB infection or evidence of currently active TB by chest x ray, residing with or frequent close contact with individual(s) with active TB.
13. Subjects receiving the following therapies within the time period described below or expected to receive any of these therapies during the study period:

    1. >9 mg/day of oral budesonide or >25 mg/day of prednisone or equivalent oral systemic corticosteroid dose within 2 weeks prior to baseline.
    2. IV, IM (parenteral), or topical (rectal) treatment of 5 ASA or corticosteroid enemas/suppositories within 2 weeks prior to baseline.
    3. Azathioprine, 6 mercaptopurine, or methotrexate within 2 weeks prior to baseline.
    4. Anti TNF inhibitors (or biosimilars thereof) as described below:

       * Infliximab within 8 weeks prior to baseline;
       * Adalimumab within 8 weeks prior to baseline;
       * Certolizumab within 8 weeks prior to baseline;
    5. Anti integrin inhibitors (eg, vedolizumab) within 8 weeks prior to baseline.
    6. Ustekinumab within 8 weeks prior to baseline.
    7. Interferon therapy within 8 weeks prior to baseline.
    8. Subjects with prior treatment with lymphocyte depleting agents/therapies within 1 year prior to baseline (eg, CamPath[alemtuzumab], alkylating agents [eg, cyclophosphamide or chlorambucil], total lymphoid irradiation, etc).
    9. Subjects who have received rituximab or other selective B lymphocyte depleting agents within 1 year prior to baseline.
    10. Subjects previously receiving leukocyte apheresis, including selective lymphocyte, monocyte, or granulocyte apheresis, or plasma exchange within 6 months prior to baseline.
    11. Other marketed immunosuppressants or biologics with immunomodulatory properties within 3 months prior to baseline.
    12. Subjects who have received other JAK inhibitors within 3 months prior to baseline.
    13. Subjects who have not responded to or have been intolerant of other JAK inhibitors.
    14. Other investigational procedures(s) or product(s), such as immunosuppressants used in transplantation (eg, mycophenolate mofetil, cyclosporine, rapamycin, or tacrolimus) or live (attenuated) vaccine within 30 days prior to baseline.

        14) Subjects with history of thrombotic event(s), including deep venous thrombosis (DVT), and known inherited conditions that predispose to hypercoagulability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (188):
- United States (51):
  - Dothan Surgery Center, Dothan, Alabama
  - Gut P.C., dba Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Brighton Surgical Center, Beverly Hills, California
  - Entertainment Medical Group, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC, Los Angeles, California
  - Stanford Medicine Outpatient Center - Digestive Health Center, Redwood City, California
  - Front Range Endoscopy Center, Colorado Springs, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Gastro Florida, Clearwater, Florida
  - West Coast Endoscopy Center, Clearwater, Florida
  - UF Health Jacksonville - Gastroenterology Emerson, Jacksonville, Florida
  - Millenia Surgery Center, Orlando, Florida
  - HMD Research LLC, Orlando, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - WestGlen Gastrointestinal Consultants, P.A., Shawnee Mission, Kansas
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Capitol Research, Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mass Eye and Ear, Longwood, Boston, Massachusetts
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Eastside Endoscopy Center, Macomb, Michigan
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical College (Colonoscopy), New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical College Investigational Pharmacy, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital (Endoscopy Suite), New York, New York
  - DiGiovanna Institute for Medical Education And Research, North Massapequa, New York
  - UNC Hospitals, Chapel Hill, North Carolina
  - UNC Hospitals Endoscopy Center at Meadowmont, Chapel Hill, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - UNC GI Procedures Hillsborough, Hillsborough, North Carolina
  - Gastroenterology Associates of the Piedmont, PA, Winston-Salem, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - Holston Valley Surgery Center, Kingsport, Tennessee
  - Vanderbilt GI Endoscopy Lab at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt Inflammatory Bowel Disease Clinic, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - First Street Hospital, Bellaire, Texas
  - First Street Surgical Center, Bellaire, Texas
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Pearland Surgery Center, Houston, Texas
  - GI Alliance, Southlake, Texas
  - Lonestar Endoscopy, LLP, Southlake, Texas
  - Texas Digestive Disease Consultants (Administrative, Regulatory), Southlake, Texas
  - Gastroenterology Associates of Northern VA, Fairfax, Virginia
  - Gastroenterology Associates of Northern Virginia, Fairfax, Virginia
  - Verity Research, Inc., Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
- Australia (4):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Mater Misericordiae Ltd, South Brisbane, Queensland
  - Ballarat Base Hospital, Ballarat, Victoria
  - Saint John of God Health Care Inc., Subiaco, Western Australia
- AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Belgium (3):
  - University Hospital Brussels, Jette
  - University Hospitals Leuven, Leuven
  - CHC MontLégia, Liége
- Javna zdravstvena ustanova Univerzitetski klinicki centar Republike Srpske,, Banja Luka, Bosnia and Herzegovina
- Winnipeg Regional Health Authority - Health Sciences Centre, Winnipeg, Winnipeg, Manitoba, Canada
- Croatia (3):
  - Klinicki Bolnicki centar Split, Zavod za gastroenterologiju, Split
  - Klinicka bolnica Dubrava Zagreb, Zagreb
  - Klinicki bolnicki centar Zagreb, Zavod za gastroenterologiju i hepatologiju, Zagreb
- Czechia (6):
  - Nemocnice Horovice, a.s., Hořovice
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - Medialpharma s.r.o., Hradec Králové
  - MUDr. GREGAR s.r.o., Olomouc
  - Nemocnice Strakonice, a.s., Interni oddeleni, Strakonice
  - Nemocnice Strakonice, a.s., Strakonice
- Georgia (3):
  - LTD "Acad. F. Todua Medical Center - LTD Research Institute of Clinical Medicine", Tbilisi
  - The First University Clinic of TSMU, Tbilisi
  - Institute of Clinical Cardiology, Ltd., Tbilisi
- Germany (3):
  - Paian MED Research GmbH, Berlin
  - Krankenhaus Waldfriede e.V.,, Berlin
  - Universitaetsklinikum Schleswig-Holstein, Kiel
- Hungary (4):
  - Bekes Megyei Kozponti Korhaz, Rethy Pal Tagkorhaz, Békéscsaba
  - Semmelweis Egyetem, II. Belgyogyaszati Klinika, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Clinfan Szolgaltato Kft., Szekszárd
- Italy (8):
  - IRCCS Saverio de Bellis, Castellana Grotte, BARI
  - A.O.Spedali Civili, Brescia, BS
  - Univ. "Magna Graecia" di Catanzaro, Catanzaro, CZ
  - ASST Monza, Monza, MB
  - Istituto Clinico Humanitas IRCCS - Sez. Autonoma di Malattie, Infiammatorie Croniche Intestinali, Rozzano, Milan
  - A.O.U. Policlinico G. Martino, Messina
  - Azienda Ospedaliera di Padova, Padua
  - Policlinico Universitario Campus Bio-Medico, Roma
- Lebanon (4):
  - American University of Beirut Medical Center, Beirut
  - Saint George Hospital University Medical Center, El Achrafiyé
  - Ain Wazein Medical Village, El Chouf
  - Hammoud Hospital University Medical Center, Saida
- Poland (35):
  - STRZEGOMSKIE CENTRUM MEDYCZNO-DIAGNOSTYCZNE Sp. z o.o., Strzegom, Lower Silesian Voivodeship
  - DC-MED Sp. z o.o. Sp.k., Swidnica, Other
  - H-T. Centrum Medyczne-Endoterapia, Tychy, Silesian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej All-Medicus, Katowice
  - ETG Kielce, Kielce
  - Indywidualna Specjalistyczna Praktyka Lekarska Maciej Zymla, Knurów
  - Szpital w Knurowie Sp. z o.o., Knurów
  - Samodzielny Publiczny Zespół Opieki Zdrowotnej, Pracownia Endoskopii, Kościan
  - Centrum Medyczne Szpital Swietej Rodziny Sp z o.o., Lodz
  - Pracownia Endoskopii Centrum Medyczne Szpital Swietej Rodziny Sp z o.o., Lodz
  - Ośrodek Badań Klinicznych Appletreeclinics, Lodz
  - SALVE, Lodz
  - Gastromed Sp. z o.o., Lublin
  - IRMED, Piotrkow Trybunalski
  - Samodzielny Szpital Wojewodzki im. M. Kopernika w Piotrkowie Trybunalskim, Piotrkow Tryunalski
  - PRZYCHODNIA SPECJALISTYCZNA MEDIC-R Clinical Research Center Spolka z ograniczona odpowiedzialnoscia, Poznan
  - Ai Centrum Medyczne Sp. Z O.O. Sp.K., Poznan
  - AM-MEDIC SP. z o.o., Poznan
  - Gabinety Lekarskie Rivermed, Poznan
  - KO-MED Centra Kliniczne, Puławy
  - Zaklad Opieki Zdrowotnej Medical Sp. z o.o., (endoscopy), Puławy
  - ENDOSKOPIA Sp. z o. o., Sopot
  - Nowe Zdrowie-CK, Kiełtucki i Wspólnicy Sp.j., Staszów
  - Twoja Przychodnia Szczecinskie Centrum Medyczne, Szczecin
  - SONOMED, Szczecin
  - Szpital Sredzki Serca Jezusowego sp. z o.o., Środa Wielkopolska
  - Centrum Zdrowia MDM, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Endoterapia PFG Sp. z o.o., Warsaw
  - Futuremeds, Wroclaw
  - Melita Medical Sp. z o.o., Wroclaw
  - Centrum Gastrologiczno Hepatologiczne, Wroclaw
  - Lexmedica, Wroclaw
  - Golden Care, Wroclaw
  - Centrum Diagnostyczno-Lecznicze Barska Sp. z o. o., Włocławek
- Russia (20):
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - SPb SBIH "City Hospital #40 of the Kurortnyi region", Saint Petersburg, Sestroretsk
  - Polyclinic Ultrasound 4D LLC, Pyatigorsk, Stavropol Kray
  - LLC "Alliance Biomedical-Ural Group", Izhevsk, Udmurt Republic
  - LLC "Alliance Biomedical-Ural Group", Izhevsk
  - LLC "Olla-Med", Moscow
  - Sechenov University on the base of Institute of Translational Medicine and Biotechnology, Moscow
  - Limited Liability Company "Medical Center SibNovoMed", Novosibirsk
  - Novosibirskiy Gastrocenter, Novosibirsk
  - Clinic at FSBEI HE "Omsk State Medical University" MoH RF, Omsk
  - LLC "New Clinic", Pyatigorsk
  - Limited Liability Company "Medical Center "Reavita Med SPb" (OOO "MC "RM SPb"), Saint Petersburg
  - Limited Liability Company "RIAT", Saint Petersburg
  - LLC "Research center Eco-Safety", Saint Petersburg
  - Limited Liability Company "RIAT SPb", Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Clinical Hospital of the Righteous, Saint Petersburg
  - Private Institution Educational Organization of Higher Education, Samara
  - Non-state Healthcare Institution 'Railway Clinical Hospital at Samara Station of Open Joint Stock, Samara
  - Limited Liability Company Medical Company "Hepatolog", Samara
  - State Budgetary Healthcare Institution of the Stavropol Region, Stavropol
- Saudi Arabia (2):
  - King AbdulAziz Medical City, Riyadh
  - King Khalid University Hospital, Riyadh
- Serbia (5):
  - Klinicko Bolnicki Centar "Bezanijska Kosa", Zemun, Beograd
  - Klinicki Centar Kragujevac, Kragujevac, Srbija
  - Opsta bolnica Subotica, Subotica, Srbija
  - Opsta Bolnica "Djordje Joanovic", Odeljenje Interno, Odsek Gastroenterologija, Zrenjanin, Srbija
  - KBC "Dr Dragisa Misovic-Dedinje", Belgrade
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, Banská Bystrica
  - ENDOMED, s.r.o., Vranov nad Topľou
- South Africa (2):
  - Wits Clinical Research Trial Site, Parktown, Gauteng
  - Dr Wright Private Practice, Claremont, Western Cape
- South Korea (3):
  - Kyungpook National University Hospital, Daegu, Korea
  - Kyung Hee University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
- Spain (5):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Universitätsspital Zürich, Zurich, Switzerland
- Tunisia (2):
  - La Rabta Hospital, Tunis
  - Habib Thameur Hospital, Tunis
- Turkey (Türkiye) (5):
  - Hacettepe Universitesi Tip Fakultesi, Ankara
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Mersin Universitesi Tip Fakultesi Hastanesi, Ic Hastaliklari, Mersin
  - Mersin Universitesi Tip Fakultesi Hastanesi, Mersin
  - Bulent Ecevit Universitesi Tip Fakultesi, Zonguldak
- Ukraine (13):
  - Regional Municipal Non-profit Enterprise "Chernivtsi Regional Clinical Hospital", Surgery Department, Chernivtsi
  - Municipal Healthcare Institution Kharkiv City Clinical Hospital #2 n.a. prof. O.O. Shalimov, Kharkiv
  - Medical Centre Medical Clinic Blagomed LLC, Kyiv
  - Medical Center "OK Clinic+" of International Institute of Clinical Trials, Kyiv
  - Medical Center "Universal clinic Oberig" of "Kapital" LLC, Gastro center, Kyiv
  - Municipal Non-profit enterprise of Kyiv Regional Council "Kyiv regional hospital", Kyiv
  - Municipal non-profit enterprise of Kyiv regional council "Kyiv regional clinical hospital", Kyiv
  - Lviv clinical hospital on Railway Transport of Health Care Center branch of PJSC Ukrainian Railway, Lviv
  - Vinnytsia City Clinical Hospital No.1, Vinnytsia
  - Private Small-Scale Enterprise Medical Center "Pulse", Vinnytsia
  - Vinnytsia Regional Clinical Hospital for War Veterans, Vinnytsia
  - Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrohov, Vinnytsia
  - Medical Center "DIACENTER"LLC, Zaporizhzhia
- Emirates Specialty Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Fensome A, Ambler CM, Arnold E, Banker ME, Brown MF, Chrencik J, Clark JD, Dowty ME, Efremov IV, Flick A, Gerstenberger BS, Gopalsamy A, Hayward MM, Hegen M, Hollingshead BD, Jussif J, Knafels JD, Limburg DC, Lin D, Lin TH, Pierce BS, Saiah E, Sharma R, Symanowicz PT, Telliez JB, Trujillo JI, Vajdos FF, Vincent F, Wan ZK, Xing L, Yang X, Yang X, Zhang L. Dual Inhibition of TYK2 and JAK1 for the Treatment of Autoimmune Diseases: Discovery of (( S)-2,2-Difluorocyclopropyl)((1 R,5 S)-3-(2-((1-methyl-1 H-pyrazol-4-yl)amino)pyrimidin-4-yl)-3,8-diazabicyclo[3.2.1]octan-8-yl)methanone (PF-06700841). J Med Chem. 2018 Oct 11;61(19):8597-8612. doi: 10.1021/acs.jmedchem.8b00917. Epub 2018 Aug 16. PMID 30113844
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of a 12-weeks induction period and a 52-weeks open label extension (OLE) period. The participants who completed induction period, entered the 52-week OLE period.
Pre-assignment Details: A total of 645 participants were screened across 26 countries of which 401 were screen failures and 244 participants were randomized in the study.
Groups:
- Induction Period: Placebo QD: Participants received placebo matched to either PF-06651600 (ritlecitinib) or PF-06700841 (brepocitinib) once daily (QD) orally for 12 weeks in induction period.
- Induction Period: Ritlecitinib 200 mg/50 mg QD: Participants received PF-06651600 (ritlecitinib) 200 milligrams (mg) QD orally for 8 weeks followed by ritlecitinib 50 mg QD orally for 4 weeks in induction period.
- Induction Period: Brepocitinib 60 mg QD: Participants received PF-06700841 (brepocitinib) 60 mg QD orally for 12 weeks in induction period.
- OLE Period: Placebo QD -> Ritlecitinib 50 mg QD: Participants who received placebo matched to ritlecitinib during the induction period were administered ritlecitinib 50 mg QD orally for 52 weeks in OLE period.
- OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD: Participants who received ritlecitinib 200 mg /50 mg QD in the induction period were administered ritlecitinib 50 mg QD for 52 weeks in OLE period.
- OLE Period: Placebo QD -> Brepocitinib 30 mg QD: Participants who received placebo matched to brepocitinib in the induction period were administered brepocitinib 30 mg QD orally for 52 weeks in OLE period.
- OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD: Participants who received brepocitinib 60 mg QD in the induction period were administered brepocitinib 30 mg QD for 52 weeks in OLE period.
Period: Induction Period (Up to 12 Weeks)
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Started | 79 | 93 | 72 | 0 | 0 | 0 | 0
Completed | 68 | 84 | 65 | 0 | 0 | 0 | 0
Not Completed | 11 | 9 | 7 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 6 | 4 | 4 | 0 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 2 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: OLE Period (Up to 52 Weeks)
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Started | 0 | 0 | 0 | 36 (Participants who received treatment in OLE period.) | 84 (Participants who received treatment in OLE period.) | 32 (Participants who received treatment in OLE period.) | 64 (Participants who received treatment in OLE period.)
Completed | 0 | 0 | 0 | 20 | 45 | 21 | 34
Not Completed | 0 | 0 | 0 | 16 | 39 | 11 | 30
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 5 | 11 | 3 | 5
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3 | 11 | 3 | 8
Not completed — No longer met eligibility criteria | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 7 | 13 | 4 | 15

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least one dose of the randomized investigational drug (ritlecitinib, brepocitinib, or placebo). Participants who received placebo in induction period were analyzed as a single reporting group.
Groups:
- Induction Period: Placebo QD: Participants received placebo matched to either PF-06651600 (ritlecitinib) or PF-06700841 (brepocitinib) QD orally for 12 weeks in induction period.
- Induction Period: Ritlecitinib 200 mg/50 mg QD: Participants received PF-06651600 (ritlecitinib) 200 mg QD orally for 8 weeks followed by ritlecitinib 50 mg QD orally for 4 weeks in induction period.
- Total: Total of all reporting groups
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD | Total
Number analyzed (Participants) | 79 | 93 | 72 | 244
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.1 (13.03) | 34.6 (10.64) | 36.5 (12.70) | 35.6 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 29 | 107
  Male | 42 | 52 | 43 | 137
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 4
  Not Hispanic or Latino | 75 | 91 | 69 | 235
  Unknown or Not Reported | 2 | 1 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 71 | 84 | 61 | 216
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Greater Than or Equal to (>=) 50 Percent (%) Reduction in Simple Endoscopic Score for Crohn's Disease (SES CD50) at Week 12: Induction Period
Description: SES CD50 was defined as 50% improvement from baseline in SES-CD. Baseline was defined as last measurement prior to first dosing on Day 1. Following bowel segments were used for calculating SES-CD scores: Ileum, right colon(C), transverse C, left C and rectum. Each segment assessed for four domains: presence of ulcers, ulcerated surface, affected surface and presence of narrowing, each scored on a scale of 0 to 3, higher scores indicated more severe condition. Presence of ulcers score: 0=none, 1=small ulcer: (0.1-0.5 centimeter[cm]), 2=Large ulcer(0.5-2 cm), 3=very large ulcer(>2 cm); ulcerated surface score: 0=none, 1=<10%, 2=10-30% and 3=>30%; affected surface score: 0=unaffected segment, 1=<50%, 2=50-75% and 3=>75%; presence of narrowing score: 0=none,1=single, can be passed, 2=multiple, can be passed and 3=cannot be passed. Total SES CD score was determined by sum of each domain score for all 5 bowel segments and ranged from 0 to 60, higher score indicating more severe disease.
Time Frame: Week 12
Population: FAS included all randomized participants who received at least one dose of the randomized investigational drug (ritlecitinib, brepocitinib, or placebo). Participants who received placebo in induction period were analyzed as a single reporting group. Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 78 | 92 | 71
Percentage of participants | 12.8 [7.1 to 19.9] | 27.2 [19.6 to 35.7] | 33.8 [25.1 to 43.1]
Statistical Analysis 1: Comparison: Induction Period: Placebo QD vs Induction Period: Ritlecitinib 200 mg/50 mg QD; Test type: Other; p = 0.0119, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 14.3, 90% CI 2-sided [4.0 to 24.5] — 90% CI was calculated using minimum (min) risk weight method (Mehrotra-Railkar 2000)
Statistical Analysis 2: Comparison: Induction Period: Placebo QD vs Induction Period: Brepocitinib 60 mg QD; Test type: Other; p = 0.0012, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 21.4, 90% CI 2-sided [10.0 to 32.9] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)

2. Primary Outcome: Number of Participants With Laboratory Test Abnormalities During OLE Period
Description: Pre-specified criteria for lab abnormalities included- hematology: hemoglobin(Hb), erythrocytes (ery),hematocrit:<0.8*lower limit of normal(LLN);reticulocytes: <0.5*LLN, >1.5*upper limit of normal(ULN); ery mean corpuscular(EMC) volume: <0.9*ULN, >1.11*ULN;EMC Hb: <0.9*LLN; platelets:>1.75*ULN; leukocytes(10^9/L): <0.6*LLN,>1.5*ULN;lymphocyte,neutrophil(10^9/L):<0.8*LLN,>1.2*ULN;basophil,eosinophil,monocyte(10^9/L):>1.2*ULN;activated partial thromboplastin time (sec): >1.1*ULN. Chemistry: bilirubin(mg/dL),aspartate aminotransferase(AT),alanine AT(units per litre)>3.0*ULN; protein, albumin(g/dL):<0.8*LLN; creatinine, triglycerides (mg/dL):>1.3*ULN; urate(mg/dL):>1.2*ULN, potassium (mEq/L):<0.9*LLN; calcium (mg/dL): <0.9*LLN,>1.1*ULN. Urinalysis: pH>8;urine,glucose,protein(mg/dl); ketones, nitrite, urine Hb(scalar):>=1. Number of participants with any lab abnormality meeting pre-specified criteria are reported.
Time Frame: From start of study intervention in OLE period up to 4 weeks after last dose of study intervention (up to 56 weeks)
Population: Safety analysis set (SAS) included all those participants who received at least one dose of the investigational drug (ritlecitinib, brepocitinib, or placebo). Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 36 | 83 | 32 | 63
Participants | 33 | 76 | 26 | 56

3. Primary Outcome: Number of Participants According to Categorization of Vital Signs During OLE Period
Description: Vital signs including blood pressure (diastolic blood pressure [DBP], systolic blood pressure [SBP], and pulse rate [PR]) were measured in a supine position using automated devices. DBP included value < 50 (millimeter of mercury [mmHg]), change >=20 (mmHg) increase and change >=20 (mmHg) decrease; SBP: value < 90 (mmHg), change >= 30 (mmHg) increase and change >= 30 (mmHg) decrease; PR: value > 120 (beats per minute [bpm]).
Time Frame: From start of study intervention in OLE period up to 4 weeks after last dose of study intervention (up to 56 weeks)
Population: SAS included all those participants who received at least one dose of the investigational drug (ritlecitinib, brepocitinib, or placebo). Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 36 | 83 | 32 | 63
Participants
  DBP; value < 50 (mmHg) | 0 | 2 | 0 | 1
  DBP; change >=20 (mmHg) increase | 4 | 6 | 2 | 6
  DBP; change >=20 (mmHg) decrease | 1 | 4 | 3 | 8
  PR; value > 120 (bpm) | 0 | 1 | 0 | 0
  SBP; value < 90 (mmHg) | 0 | 2 | 0 | 1
  SBP; change >= 30 (mmHg) increase | 1 | 2 | 0 | 5
  SBP; change >= 30 (mmHg) decrease | 3 | 0 | 3 | 2

4. Primary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiogram Findings During OLE Period
Description: Single twelve lead ECGs were obtained using an automated ECG machine after participant had rested quietly for at least 10 minutes in a supine position. QTc prolongations were defined as a QTc >=480 milli second (msec) or an absolute change in QTc greater than (>) 60 msec. Clinically significant ECG findings were determined by the investigator.
Time Frame: From start of study intervention in OLE period up to 4 weeks after last dose of study intervention (up to 56 weeks)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 23 | 50 | 21 | 40
Participants | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During OLE Period
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a study intervention; the event need not necessarily have a causal relationship with the treatment or usage. An AE was considered TEAE to a given treatment if the event started during the effective duration of treatment regardless of whether a similar event of equal or greater severity existed in the baseline period.
Time Frame: From start of study intervention in OLE period up to 4 weeks after last dose of study intervention (up to 56 weeks)
Population: SAS included all those participants who received at least one dose of the investigational drug (ritlecitinib, brepocitinib, or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 36 | 84 | 32 | 64
Participants | 32 | 58 | 25 | 54

6. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAE) During OLE Period
Description: A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions) or resulted in congenital anomaly/birth defect or was considered an important medical event. An SAE was considered as TESAE if the event started during the effective duration of treatment regardless of whether a similar event of equal or greater severity existed in the baseline period.
Time Frame: From start of study intervention in OLE period up to 4 weeks after last dose of study intervention (up to 56 weeks)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 36 | 84 | 32 | 64
Participants | 6 | 10 | 5 | 16

7. Primary Outcome: Number of Participants With Discontinuations Due to Adverse Events During OLE Period
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention; the event need not necessarily have a causal relationship with the treatment or usage. Discontinuations from study due to TEAEs were defined as participants with an AE record indicating the AE caused permanent discontinuation from the study but action taken with study treatment was not drug withdrawn. Permanent discontinuations from any study intervention due to TEAEs were defined as participants with an AE record indicating that action taken with study treatment was drug withdrawn. In this outcome measure number of participants with discontinuation from study due to AEs and permanent discontinuation from study intervention due to AEs are reported.
Time Frame: From start of study intervention in OLE period up to 4 weeks after last dose of study intervention (up to 56 weeks)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 36 | 84 | 32 | 64
Participants
  Discontinuation from study due to TEAEs | 0 | 1 | 0 | 0
  Permanent discontinuation from any study intervention due to TEAEs | 7 | 13 | 4 | 15

8. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities During Induction Period
Description: Pre-specified criteria for lab abnormalities included- hematology: hemoglobin, erythrocytes, hematocrit:<0.8*LLN; reticulocytes: <0.5*LLN, >1.5*ULN; EMC volume: <0.9*ULN, >1.11*ULN;EMC Hb: <0.9*LLN; platelets:>1.75*ULN; leukocytes(10^9/L): <0.6*LLN, >1.5*ULN; lymphocyte, neutrophil(10^9/L):<0.8*LLN, >1.2*ULN; basophil, eosinophil, monocyte(10^9/L):>1.2*ULN; activated partial thromboplastin time (sec): >1.1*ULN. Chemistry: bilirubin(mg/dL),aspartate aminotransferase(AT),alanine AT(units per litre)>3.0*ULN; protein, albumin(g/dL):<0.8*LLN; creatinine, triglycerides (mg/dL):>1.3*ULN; urate(mg/dL):>1.2*ULN, potassium (mEq/L):<0.9*LLN; calcium (mg/dL): <0.9*LLN,>1.1*ULN. Urinalysis: pH>8; urine, glucose, protein(mg/dl); ketones, nitrite, urine Hb(scalar):>=1. Number of participants with any lab abnormality meeting pre-specified criteria are reported.
Time Frame: From start of study intervention on Day 1 up to Week 12
Population: SAS included all those participants who received at least one dose of the investigational drug (ritlecitinib, brepocitinib, or placebo). Participants who received placebo in induction period were analyzed as a single reporting group. Here "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 78 | 92 | 72
Participants | 67 | 72 | 61

9. Secondary Outcome: Number of Participants According to Categorization of Vital Signs During Induction Period
Description: Vital signs including blood pressure (diastolic blood pressure [DBP], systolic blood pressure [SBP], and pulse rate [PR]) were measured in a supine position using automated devices. DBP included value < 50 (mmHg), change >=20 (mmHg) increase and change >=20 (mmHg) decrease; SBP: value < 90 (mmHg), change >= 30 (mmHg) increase and PR: value > 120 (bpm).
Time Frame: From start of study intervention on Day 1 up to Week 12
Population: SAS included all those participants who received at least one dose of the investigational drug (ritlecitinib, brepocitinib, or placebo). Participants who received placebo in induction period were analyzed as a single reporting group. Here, 'Number Analyzed' signifies number of participants evaluable for specific rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 79 | 93 | 72
Participants
  Diastolic blood pressure; value < 50 (mmHg) | 1 | 0 | 0
  Diastolic blood pressure; change >=20 (mmHg) increase: number analyzed (Participants) | 78 | 92 | 72
  Diastolic blood pressure; change >=20 (mmHg) increase | 4 | 2 | 4
  Diastolic blood pressure; change >=20 (mmHg) decrease: number analyzed (Participants) | 78 | 92 | 72
  Diastolic blood pressure; change >=20 (mmHg) decrease | 4 | 2 | 4
  Pulse rate; value > 120 (bpm) | 4 | 1 | 0
  Systolic blood pressure; value < 90 (mmHg) | 0 | 3 | 0
  Systolic blood pressure; change >= 30 (mmHg) increase: number analyzed (Participants) | 78 | 92 | 72
  Systolic blood pressure; change >= 30 (mmHg) increase | 3 | 2 | 7
  Systolic blood pressure; change >= 30 (mmHg) decrease: number analyzed (Participants) | 78 | 92 | 72
  Systolic blood pressure; change >= 30 (mmHg) decrease | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormal Clinically Significant Electrocardiogram Findings During Induction Period
Description: Single twelve lead ECGs were obtained using an automated ECG machine after participant had rested quietly for at least 10 minutes in a supine position. QTc prolongations were defined as a QTc greater than or equal to (>=)480 milli second (msec) or an absolute change in QTc greater than (>)60 msec. Clinically significant ECG findings were determined by the investigator.
Time Frame: From start of study intervention on Day 1 up to Week 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 68 | 83 | 63
Participants | 1 | 0 | 0

11. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) During Induction Period
Description: An AE was any untoward medical occurrence in a study participant administered a study intervention; the event need not necessarily have a causal relationship with the treatment or usage. An AE was considered TEAE to a given treatment if the event started during the effective duration of treatment regardless of whether a similar event of equal or greater severity existed in the baseline period.
Time Frame: From start of study intervention on Day 1 up to Week 12
Population: SAS included all those participants who received at least one dose of the investigational drug (ritlecitinib, brepocitinib, or placebo). Participants who received placebo in induction period were analyzed as a single reporting group.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 79 | 93 | 72
Participants | 51 | 46 | 49

12. Secondary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAE) During Induction Period
Description: A SAE was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions) or resulted in congenital anomaly/birth defect or was considered an important medical event. An SAE was considered as TESAE if the event started during the effective duration of treatment regardless of whether a similar event of equal or greater severity existed in the baseline period.
Time Frame: From start of study intervention on Day 1 up to Week 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 79 | 93 | 72
Participants | 6 | 4 | 4

13. Secondary Outcome: Number of Participants Discontinuation Due to Adverse Events During Induction Period
Description: as for outcome 7
Time Frame: From start of study intervention on Day 1 up to Week 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 79 | 93 | 72
Participants
  Discontinuations from study due to TEAEs | 0 | 1 | 0
  Permanent discontinuations from any study intervention due to TEAEs | 6 | 4 | 4

14. Secondary Outcome: Number of Participants With Serious Infections During Induction Period
Description: Participants were monitored for development of any infection (viral, bacterial and fungal). Serious infections were treated infections that required parenteral antimicrobial therapy and were present with positive pre-treatment culture and required hospitalization for treatment/met other criteria that required the infection to be classified as SAE. An SAE was any untoward medical occurrence at any dose that: resulted in death; is life-threatening; requires inpatient hospitalization/prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity/results in congenital anomaly/birth defect. Treated infections were infections that required antimicrobial therapy by any route of administration/required any surgical intervention (e.g., incision and drainage).
Time Frame: From start of study intervention on Day 1 up to Week 12
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 79 | 93 | 72
Participants | 0 | 1 | 2

15. Secondary Outcome: Percentage of Participants Who Achieved Clinically Meaningful Endoscopic Improvement (CMEI) (Reduction of >=3 Points From Baseline in SES-CD Score) at Week 12: Induction Period
Description: CMEI was defined as reduction of >=3 points from baseline in SES-CD score as assessed by centrally read SES-CD score. Baseline: last measurement prior to first dosing on Day1. Following bowel segments were used for calculating SES-CD scores: Ileum, right C, transverse C, left C and rectum. Each segment assessed for 4 domains: presence of ulcers, ulcerated surface, affected surface and presence of narrowing, each scored on scale of 0-3, higher scores indicated more severe condition. Presence of ulcers score: 0=none,1=small ulcer: (0.1-0.5cm),2=Large ulcer(0.5-2cm),3=very large ulcer(>2cm); ulcerated surface score: 0=none,1=<10%,2=10-30% and 3=>30%; affected surface score: 0=unaffected segment, 1=<50%, 2=50-75% and 3=>75%; presence of narrowing score: 0=none,1=single, can be passed, 2=multiple, can be passed and 3=cannot be passed. Total SES CD score was determined by sum of each domain score for all 5 bowel segments and ranged from 0 to 60, higher score indicating more severe disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 78 | 92 | 71
Percentage of participants | 29.5 [21.7 to 38.9] | 42.4 [34.2 to 51.5] | 57.7 [47.6 to 67.2]
Statistical Analysis 1: Comparison: Induction Period: Placebo QD vs Induction Period: Ritlecitinib 200 mg/50 mg QD; Test type: Other; p = 0.0390, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 13.3, 90% CI 2-sided [1.0 to 25.7] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)
Statistical Analysis 2: Comparison: Induction Period: Placebo QD vs Induction Period: Brepocitinib 60 mg QD; Test type: Other; p = 0.0001, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 29.7, 90% CI 2-sided [17.2 to 42.2] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)

16. Secondary Outcome: Mean Change From Baseline in SES-CD Score at Week 12: Induction Period
Description: Mean change from baseline in SES-CD score at Week 12 analyzed using analysis of covariance(ANCOVA)model with treatment,baseline disease activity/extent as factors, baseline SES CD score as covariate. Baseline=last measurement prior to first dosing on Day 1. Following bowel segments used for calculating SES-CD scores: Ileum,right C,transverse C,left C,rectum. Each segment assessed for four domains:presence of ulcers, ulcerated surface, affected surface,presence of narrowing, each score on a scale of 0-3,higher scores=more severe condition. Presence of ulcers score:0=none,1=small ulcer:(0.1-0.5cm),2=large ulcer(0.5-2cm),3=very large ulcer(>2 cm);ulcerated surface score:0=none,1=<10%,2=10-30%,3=>30%;affected surface score:0=unaffected segment,1=<50%, 2=50-75%,3=>75%;presence of narrowing score:0=none,1=single,can be passed,2=multiple can be passed,3=cannot be passed. Total SES CD score=sum of each domain score for all 5 bowel segments,range from 0 to 60,higher score =more severe disease.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Units on a scale
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 68 | 82 | 63
Units on a scale | -0.1 [-1.32 to 1.12] | -3.1 [-4.22 to -2.02] | -5.0 [-6.36 to -3.72]
Statistical Analysis 1: Comparison: Induction Period: Placebo QD vs Induction Period: Ritlecitinib 200 mg/50 mg QD; Test type: Other; p = 0.0007, ANCOVA; The ANCOVA model included treatment and baseline disease activity/extent as factors, and baseline SES-CD score as a covariate; LS mean difference = -3.0, 90% CI 2-sided [-4.55 to -1.48]
Statistical Analysis 2: Comparison: Induction Period: Placebo QD vs Induction Period: Brepocitinib 60 mg QD; Test type: Other; p < .0001, ANCOVA; [statistical method as in outcome 16, analysis 1]; LS mean difference = -4.9, 90% CI 2-sided [-6.62 to -3.26]

17. Secondary Outcome: Percentage of Participants Achieving >=25% Reduction in SES-CD From Baseline (SES-CD 25) at Week 12: Induction Period
Description: SES CD25 was defined as >=25% improvement from baseline in SES CD. Baseline was defined as the last measurement prior to first dosing on Day 1. Following bowel segments were used for calculating SES-CD scores: Ileum, right C, transverse C, left C and rectum. Each segment assessed for four domains: presence of ulcers, ulcerated surface, affected surface and presence of narrowing, each scored on a scale of 0 to 3, higher scores indicated more severe condition. Presence of ulcers score: 0=none, 1=small ulcer: (0.1-0.5 centimeter[cm]), 2=Large ulcer(0.5-2 cm), 3=very large ulcer(>2 cm); ulcerated surface score: 0=none, 1=<10%, 2=10-30% and 3=>30%; affected surface score: 0=unaffected segment, 1=<50%, 2=50-75% and 3=>75%; presence of narrowing score: 0=none,1=single, can be passed, 2=multiple, can be passed and 3=cannot be passed. Total SES CD score was determined by sum of each domain score for all 5 bowel segments and ranged from 0 to 60, higher score indicating more severe disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 78 | 92 | 71
Percentage of participants | 25.6 [17.7 to 34.3] | 39.1 [30.6 to 47.4] | 56.3 [46.2 to 66.4]
Statistical Analysis 1: Comparison: Induction Period: Placebo QD vs Induction Period: Ritlecitinib 200 mg/50 mg QD; Test type: Other; p = 0.0279, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 13.9, 90% CI 2-sided [2.1 to 25.6] — 90% CI was calculated using using minimum risk weight method (Mehrotra-Railkar, 2000)
Statistical Analysis 2: Comparison: Induction Period: Placebo QD vs Induction Period: Brepocitinib 60 mg QD; Test type: Other; p < .0001, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 31.5, 90% CI 2-sided [19.1 to 43.9] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)

18. Secondary Outcome: Percentage of Participants Achieving Endoscopic Remission (SES-CD Score of <= 2) at Week 12: Induction Period
Description: Endoscopic remission was defined as SES-CD score of <= 2. Following bowel segments were used for calculating SES-CD scores: Ileum, right colon(C), transverse C, left C and rectum. Each segment assessed for four domains: presence of ulcers, ulcerated surface, affected surface and presence of narrowing, each scored on a scale of 0 to 3, higher scores indicated more severe condition. Presence of ulcers score: 0=none, 1=small ulcer: (0.1-0.5 centimeter[cm]), 2=Large ulcer(0.5-2 cm), 3=very large ulcer(>2 cm); ulcerated surface score: 0=none, 1=<10%, 2=10-30% and 3=>30%; affected surface score: 0=unaffected segment, 1=<50%, 2=50-75% and 3=>75%; presence of narrowing score: 0=none,1=single, can be passed, 2=multiple, can be passed and 3=cannot be passed. Total SES CD score was determined by sum of each domain score for all 5 bowel segments and ranged from 0 to 60, higher score indicating more severe disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 78 | 92 | 71
Percentage of participants | 5.1 [2.3 to 11.2] | 7.6 [4.0 to 13.2] | 12.7 [7.2 to 20.8]
Statistical Analysis 1: Comparison: Induction Period: Placebo QD vs Induction Period: Ritlecitinib 200 mg/50 mg QD; Test type: Other; p = 0.2922, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 2.5, 90% CI 2-sided [-4.3 to 9.3] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)
Statistical Analysis 2: Comparison: Induction Period: Placebo QD vs Induction Period: Brepocitinib 60 mg QD; Test type: Other; p = 0.0449, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 7.4, 90% CI 2-sided [-0.4 to 15.2] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)

19. Secondary Outcome: Percentage of Participants Achieving Mucosal Healing at Week 12: Induction Period
Description: Mucosal healing was defined as complete absence of ulcers.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD
Number analyzed (Participants) | 78 | 92 | 71
Percentage of participants | 5.1 [2.3 to 11.2] | 10.9 [6.1 to 17.7] | 16.9 [10.1 to 25.8]
Statistical Analysis 1: Comparison: Induction Period: Placebo QD vs Induction Period: Ritlecitinib 200 mg/50 mg QD; Test type: Other; p = 0.0998, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 5.8, 90% CI 2-sided [-1.6 to 13.3] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)
Statistical Analysis 2: Comparison: Induction Period: Placebo QD vs Induction Period: Brepocitinib 60 mg QD; Test type: Other; p = 0.0111, Min risk weight method(Mehrotra-Railkar); Percentage risk difference = 11.8, 90% CI 2-sided [2.8 to 20.9] — 90% CI was calculated using minimum risk weight method (Mehrotra-Railkar, 2000)

20. Secondary Outcome: Percentage of Participants Achieving CMEI at Week 64 Among Participants Who Achieved CMEI Response at Week 12 (Baseline of OLE Period): OLE Period
Description: CMEI was defined as reduction of >=3 points from baseline as assessed by centrally read SES CD score. Baseline: last measurement prior to first dosing on Day 1 of Week 12. Following bowel segments were used for calculating SES-CD scores: Ileum, right C, transverse C, left C and rectum. Each segment assessed for four domains: presence of ulcers, ulcerated surface, affected surface and presence of narrowing, each scored on scale of 0-3, higher scores indicated more severe condition. Presence of ulcers score: 0=none,1=small ulcer: (0.1-0.5 cm),2=Large ulcer(0.5-2 cm),3=very large ulcer(>2 cm); ulcerated surface score: 0=none,1=<10%, 2=10-30% and 3=>30%; affected surface score: 0=unaffected segment, 1=<50%, 2=50-75% and 3=>75%; presence of narrowing score: 0=none,1=single, can be passed, 2=multiple, can be passed and 3=cannot be passed. Total SES CD score was determined by sum of each domain score for all 5 bowel segments and ranged from 0-60, higher score indicating more severe disease.
Time Frame: Week 64 (Week 52 of OLE period)
Population: FAS included all randomized participants who received at least one dose of the randomized investigational drug (ritlecitinib, brepocitinib, or placebo). Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 11 | 34 | 11 | 38
Percentage of participants | 27.3 [10.5 to 56.4] | 44.1 [30.7 to 59.5] | 54.5 [30.2 to 80.0] | 42.1 [28.5 to 56.7]

21. Secondary Outcome: Percentage of Participants Achieving SES CD 25 and SES CD 50 at Week 64 Among Participants Who Achieved SES CD 25 and SES CD 50 at Week 12 (Baseline of OLE Period): OLE Period
Description: SES CD50 and SES CD25: 50% and 25% improvement from baseline, respectively. Baseline: last measurement prior to first dosing on Day 1 of Week 12. Following bowel segments were used for calculating SES-CD scores: Ileum, right C, transverse C, left C and rectum. Each segment assessed for four domains: presence of ulcers, ulcerated surface, affected surface and presence of narrowing, each scored on a scale of 0 to 3, higher scores indicated more severe condition. Presence of ulcers score: 0=none, 1=small ulcer: (0.1-0.5 cm), 2=Large ulcer(0.5-2 cm), 3=very large ulcer(>2 cm); ulcerated surface score: 0=none, 1=<10%, 2=10-30% and 3=>30%; affected surface score: 0=unaffected segment, 1=<50%, 2=50-75% and 3=>75%; presence of narrowing score: 0=none,1=single, can be passed, 2=multiple, can be passed and 3=cannot be passed. Total SES CD score was determined by sum of each domain score for all 5 bowel segments and ranged from 0 to 60, higher score indicating more severe disease.
Time Frame: Week 64 (Week 52 of OLE period)
Population: FAS included all randomized participants who received at least one dose of the randomized investigational drug (ritlecitinib, brepocitinib, or placebo). Here "Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed"=participants evaluable for specified rows.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
Number analyzed (Participants) | 8 | 31 | 11 | 38
Percentage of participants
  SES-CD 25 | 25.0 [6.9 to 58.2] | 41.9 [26.9 to 57.9] | 54.5 [30.2 to 80.0] | 42.1 [28.5 to 56.7]
  SES-CD 50: number analyzed (Participants) | 4 | 22 | 6 | 22
  SES-CD 50 | 25.0 [2.6 to 68.0] | 36.4 [19.6 to 55.6] | 50.0 [20.1 to 79.9] | 36.4 [19.6 to 55.6]

ADVERSE EVENTS:
Time Frame: Induction Period: From start of study intervention on Day 1 up to Week 12 (for a maximum duration of 12 weeks); OLE Period: From start of study intervention in OLE period (Week 12) up to 4 weeks after last dose of study intervention on Week 64 (for a maximum duration of 56 weeks)
Description: Same event may appear as both non-SAE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and non-serious in another participants, or one participant may have experienced both serious and non-serious event during the study.
Arm/Group | Induction Period: Placebo QD | Induction Period: Ritlecitinib 200 mg/50 mg QD | Induction Period: Brepocitinib 60 mg QD | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD | OLE Period: Placebo QD -> Brepocitinib 30 mg QD | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/93 | 0/72 | 0/36 | 0/84 | 0/32 | 0/64
Serious Adverse Events (participants affected / at risk) | 6/79 | 4/93 | 4/72 | 6/36 | 10/84 | 5/32 | 16/64
Other Adverse Events (participants affected / at risk) | 20/79 | 20/93 | 17/72 | 29/36 | 34/84 | 19/32 | 31/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Placebo QD (N=79) | Induction Period: Ritlecitinib 200 mg/50 mg QD (N=93) | Induction Period: Brepocitinib 60 mg QD (N=72) | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD (N=36) | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD (N=84) | OLE Period: Placebo QD -> Brepocitinib 30 mg QD (N=32) | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD (N=64)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 5 | 2 | 0 | 3 | 5 | 3 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bartholin's abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mesenteric abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction Period: Placebo QD (N=79) | Induction Period: Ritlecitinib 200 mg/50 mg QD (N=93) | Induction Period: Brepocitinib 60 mg QD (N=72) | OLE Period: Placebo QD -> Ritlecitinib 50 mg QD (N=36) | OLE Period: Ritlecitinib 200 mg/50 mg QD -> Ritlecitinib 50 mg QD (N=84) | OLE Period: Placebo QD -> Brepocitinib 30 mg QD (N=32) | OLE Period: Brepocitinib 60 mg QD -> Brepocitinib 30 mg QD (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 4 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 4 | 4 | 5 | 4 | 6
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 4 | 2 | 2 | 4 | 9 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 3
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 3 | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 0 | 1 | 3 | 2 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
SARS-CoV-2 test positive (Investigations) | 3 | 6 | 1 | 6 | 4 | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 2 | 2 | 1 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 5 | 1 | 1 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 4 | 1 | 1 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03395184/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03395184/SAP_001.pdf